CLINICAL TRIAL: NCT00898664
Title: Genetic Analysis of Head and Neck Squamous Cell Carcinoma
Brief Title: DNA Analysis of Tissue Samples From Patients With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC HN 0625; VU-VICC-HN-0625; VU-VICC-IRB-060462
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; stage I squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; salivary gland squamous cell carcinoma; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Cytogenetic Analysis; Gene Expression Profiling; Polymerase Chain Reaction; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Assess common genetic mutations in tumor and germline DNAs from HNSCCs and search for viral DNAs and relate this information to demographics, tumor characteristics and patient prognosis.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: cytogenetic analysis
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at DNA in tissue samples from patients with head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess common genetic mutations in tumor and germline DNA samples from patients with head and neck squamous cell carcinoma (HNSCC).
* Search for viral DNAs and relate this information to demographics, tumor characteristics, and patient prognosis.
* Search for novel viral sequences and cancer-associated gene mutations in young nonsmoking HNSCC patients and in other distinct head and neck cancers.
* Determine tumor suppressor gene mutations in HNSCC patients and relate this information to gene expression data.
* Validate gene expression information using independent techniques such as real-time PCR on expressed sequences and immunohistochemistry.

OUTLINE: Genetic mutation analysis and gene expression studies are performed on tissue samples from patients with head and neck squamous cell carcinoma. Techniques used include real time-PCR and immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Patient with head and neck squamous cell carcinoma (HNSCC) enrolled in the Head and Neck Tissue Repository

  * Sufficient biological material collected to perform study tests
* Historical material available from excess tissues at the Vanderbilt Pathology Department

Exclusion Criteria:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nonsmoking patients less than 40 years of age at first diagnosis of HNSCC.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2006-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Assess common genetic mutations in tumor and germline DNA samples | Upon collection of final patient data
Viral DNAs related to demographics, tumor characteristics, and patient prognosis | Upon collection of final patient data
Novel viral sequences and cancer-associated gene mutations in young nonsmoking patients with head and neck squamous cell carcinoma and in other distinct head and neck cancers | Upon collection of final patient data
Tumor suppressor gene mutations related to gene expression data | upon collection of final patient data
Validation of gene expression information using independent techniques such as real-time PCR on expressed sequences and immunohistochemistry | upon collection of final patient data

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Murphy, MD, Study Chair — Vanderbilt-Ingram Cancer Center